CLINICAL TRIAL: NCT04886128
Title: Improving Diagnostic Accuracy for Acute Heart Failure
Acronym: INDICATE-HF
Status: Active, not recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Wayne State University (Other)
Responsible Party: Principal Investigator, Deepak Gupta, Assistant Professor, Director, Vanderbilt University Medical Center
Other Study IDs: 210941
Record Dates: First submitted 2021-05-04; First posted 2021-05-13 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Acute Heart Failure; Dyspnea; Dyspnea; Cardiac
Keywords: heart failure; acute heart failure
MeSH Terms: conditions — Dyspnea; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma, serum, whole blood, and urine samples will be retained. For the primary aims, plasma will be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Aim 1/Outcome 1: Secondary analysis of frozen plasma samples from the existing STRATIFY cohort of patients with and without acute heart failure presenting to emergency departments. n= ~900
- Aim2/Outcome 2: Secondary analysis of frozen plasma samples from the existing EMROC cohort of patients with and without acute heart failure presenting to emergency departments. n= ~900
- Aim 3/Outcome 3: Prospective recruitment of approximately 1000 patients with and w/o acute heart failure presenting to emergency departments.

SUMMARY:
Acute heart failure is a common reason for emergency department visits and hospitalization, but the diagnosis can be challenging because of non-specific symptoms and signs. The current diagnostic approach to acute heart failure has modest accuracy, leading to delayed diagnosis and treatment, which associate with worse prognosis. Prior work suggests diagnostic accuracy can be improved with the addition of multiple circulating biomarkers discovered through proteomics, and this study will derive and validate a multi-marker model to improve diagnostic accuracy for acute heart failure in the emergency department.

DETAILED DESCRIPTION:
Acute heart failure (HF) is highly morbid, lethal, and costly. It is a difficult diagnosis to make given its symptoms and signs overlap with other cardiac and non-cardiac conditions. In the emergency department (ED), misdiagnosis of acute HF is common and associated with adverse outcomes. Biomarker testing can facilitate accurate diagnosis; however, natriuretic peptides (NP) are the only guideline recommend biomarker of HF for diagnostic testing, and are better for ruling-out, rather than ruling-in, acute HF. Even with NP testing, in contemporary clinical practice misdiagnosis of acute HF still occurs in 10 to 45% of patients presenting to the ED with dyspnea. Clinical prediction models including multiple biomarkers hold promise for improving diagnostic accuracy. The few prior studies investigating a multiple biomarker approach for diagnosing acute HF were limited by constraint to highly correlated markers from known biologic pathways, relatively small sample sizes, lack of inclusion of all a priori selected biomarkers into a single model, and absence of validation cohorts. The current study is designed to address these limitations. Recent advances in "omics" enable novel biomarker discovery on a larger scale and investigations less "biased" by existing knowledge. The overarching hypothesis of this study is that a multi-marker model incorporating novel proteins discovered with plasma proteomics improves diagnostic accuracy for acute HF. In a preliminary proof of concept study plasma proteomics was utilized to discover a multi-marker panel of 21 biomarkers which improved diagnostic accuracy for acute HF beyond current clinical practice using clinical data and NP levels. These promising preliminary data motivate broader discovery in a larger sample size with subsequent derivation and validation of a multi-marker model for diagnosing acute HF in independent samples of adequate size. The specific aims of this study are to: 1) discover a multi-marker panel of 21 biomarkers to improve diagnostic accuracy for acute HF, 2) derive a model for diagnosing acute HF incorporating the 21-biomarker panel, and 3) test performance of the multi-marker model in a prospective validation cohort. In aim 1, existing plasma samples from ~900 patients will be used to assay 925 proteins to discover a smaller set of novel biomarkers most strongly associated with an adjudicated acute HF diagnosis. In aim 2, an existing prospective observational cohort, EMROC-AHF, will be utilized to derive the multi-marker model in ~900 patients who presented to the ED with acute dyspnea. In aim 3, from four EDs in Detroit, MI and Nashville, TN a new sample will prospectively recruit ~1,000 patients presenting with acute dyspnea and adjudicate the presence of acute HF by cardiologist panel review. Given the burden of HF, the frequency of inaccurate diagnosis and its adverse consequences, this study will address a significant unmet need by improving diagnostic accuracy for acute HF.

ELIGIBILITY:
For enrollment into the prospective cohort for Outcome 3.

Inclusion Criteria:

1. Willing to adhere to the study protocol
2. Able to provide written consent
3. English or Spanish speaking
4. Adult, defined as 18 years or older
5. Primary reason for presentation to the ED is dyspnea
6. ED physician is considering a diagnosis of HF, defined by ordering a NP test and/or a chest x-ray

Exclusion Criteria:

1. History of end-stage renal disease for which hemodialysis is needed
2. Dyspnea due to primary presentation of an acute coronary syndrome or trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (18 years or older) presenting with the chief complaint of dyspnea and in whom the ED physician is considering the diagnosis of acute HF, based on an order for measurement of NP levels (either BNP or NT-proBNP) or a chest x-ray will be included. Patients whose dyspnea is due to trauma, those who are on chronic hemodialysis, and patients whose primary presentation is consistent with acute coronary syndrome will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 2800 (Estimated)
Dates: Start 2021-08-31 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Biomarker Discovery | Enrollment
  Define the multi-marker panel of 21 proteins that may improve diagnostic accuracy for acute heart failure
Model derivation for diagnosing acute HF | Enrollment
  derive a model for diagnosing acute HF incorporating the 21-biomarker panel from outcome 1
Model validation for diagnosing acute HF | Enrollment
  test performance of the multi-marker model (from outcome 2) in a prospective validation cohort

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Gupta, MD, MSCI, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided